CLINICAL TRIAL: NCT02691689
Title: Prospective, Monocentric Pilot Study for the Identification of Known or Novel Genes Associated With Development of Pulmonary Arterial Hypertension in Patients With Congenital Shunt Lesions
Brief Title: Genes Associated With Development of Pulmonary Arterial Hypertension in Patients With Congenital Shunt Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Werner Budts, Werner Budts, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S57936
Record Dates: First submitted 2016-02-17; First posted 2016-02-25 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Heart Defects, Congenital; Pulmonary Arterial Hypertension; Genetic Testing
MeSH Terms: conditions — Heart Defects, Congenital; Pulmonary Arterial Hypertension | interventions — Genetic Testing

ARMS (1):
- Patients with ASD or VSD and PAH (Other)
  Interventions: Other: Genetic testing

INTERVENTIONS:
Other: Genetic testing — Genetic testing by DNA sequencing on blood samples after DNA extraction

SUMMARY:
Pulmonary arterial hypertension (PAH) in patients with congenital heart disease (CHD) is associated with considerable morbidity and even mortality.

Next to environmental risk factors, the investigators believe that there is an important role of genetic predisposition to develop PAH in CHD. There often is a discrepancy between the severity of PAH and the CHD, where it is useful to screen for PAH gene mutations. The investigators hypothesize that the genotype is partly responsible for the phenotypic variability in patients with congenital shunt lesions, where some develop PAH and others do not. If a genetic predisposition for PAH in CHD could be identified, then genetic screening could be a useful additional tool for early detection of patients at risk of pulmonary vascular disease and PAH development, with new opportunities for prevention or early treatment.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) in patients with congenital heart disease (CHD) usually develops secondary to chronic volume overload of the pulmonary circulation following left to right shunt. This overload leads to elevated pulmonary artery pressure (PAP) and later to increased pulmonary vascular resistance. This causes pressure overload in the right heart, and thereby right ventricular and right atrial dysfunction, which may implicate considerable morbidity and even mortality.

Since PAH nowadays is mostly detected when symptoms occur and PAP are elevated, the disease already evolved to an advanced (partially irreversible) stage and treatment is often initiated too late.

Next to environmental risk factors, the investigators believe that there is an important role of genetic predisposition to develop PAH in CHD. In the past, certain genes have been identified that play a role in the development of atrial septal defect (ASD). There are also a lot of genes identified that play a role in PAH. Until now, not many research groups have studied a genetic link between CHD and PAH development. But it becomes more and more clear that there often is a discrepancy between the severity of PAH and the CHD, where it is useful to screen for PAH gene mutations. The investigators hypothesize that mutations in some of these known PAH genes or in other, still unidentified, genes are partly responsible for the phenotypic variability in patients with congenital shunt lesions, where some develop PAH and others do not. If a genetic predisposition for PAH in CHD could be identified, then genetic screening could be a useful additional tool for early detection of patients at risk of pulmonary vascular disease and PAH development, with new opportunities for prevention or early treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of secundum atrial septal defect (ASD) or ventricular septal defect (VSD), with or without repair
* Development of PAH, defined as mean PAP ≥ 25 mmHg by right heart catheterization, in combination with a pulmonary wedge pressure of ≤ 15 mmHg and a PVR (pulmonary vascular resistance) of > 3 Wood units
* Preferably, families with congenital shunt lesions (at least three family members affected with ASD or VSD) will be considered for inclusion

Exclusion Criteria:

* Other congenital heart disease
* Mental retardation
* Dysmorphic characteristics
* Chronic lung disease or total lung capacity < 80% of predicted value
* History of pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2015-11; Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Presence of pathogenic mutations in PAH or ASD genes | 18 months
  * In a first step, known PAH genes (BMPR2, ALK1 and endoglin) will be screened for mutations.
  * In a second step, known ASD genes will be screened.
  * If step 1 and 2 remain negative, exome sequencing will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Budts, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium